CLINICAL TRIAL: NCT02080052
Title: Robot-Assisted MRI-Guided Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: J1163; 1RC1EB010936-01 (NIH); NA_00025078 (Other: JHMIRB)
Record Dates: First submitted 2014-02-06; First posted 2014-03-06 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Robot-assisted prostate biopsy (Experimental)
  Interventions: Device: Robot-assisted prostate biopsy

INTERVENTIONS:
Device: Robot-assisted prostate biopsy

SUMMARY:
Prostate biopsies are commonly performed freehanded under transrectal ultrasound guidance (TRUS). Due to the manual approach and the limitations of the ultrasound imager, the procedure has high false-negative rates. This represents a daily problem for urologists managing the disease, creates uncertainty and emotional stress for patients, and initiates a cascade of repeat testing and biopsies which also burden the investigators healthcare system.

The investigators believe that prostate biopsy can be improved by using a new biopsy paradigm. The investigators plan to perform MRI-guided prostate biopsies with robot-assistance for orienting a needle-guide through which the biopsy is taken. The combination of MRI and robotic precision is expected to improve prostate biopsy sensitivity compared to regular TRUS biopsies.

The study is a Pilot clinical trial on 5 patients to primarily assess feasibility and safety. The needle-guide robot is an investigational device developed in their Urology Robotics Laboratory.

DETAILED DESCRIPTION:
While prostate cancer is the most common non-dermatologic malignancy among men in the US, it is frequently indolent and may not require radical therapy, i.e. radical prostatectomy or external beam radiotherapy. There has been increased interest in conservative approaches to low risk disease, including both active surveillance and focal therapy. Both of these approaches require accurate mapping of the prostate to allow for reproducible access to diseased portions of the gland, for biopsy or treatment purposes. Magnetic resonance imaging (MRI) has been increasingly utilized for prostate cancer staging and is considered the most accurate technique available for imaging prostate cancer. Furthermore there is increasing concern about the use of freehand transrectal ultrasound (TRUS) and needle biopsying in terms of reproducibility and accuracy in mapping disease. With systematic TRUS-guided biopsy the sensitivity of the test is low (33%-44%) and yields high false-negative rates (23%) [1, 2].

The investigators hypothesize that the integration of a novel robotic device for assisting MRI-guided prostate biopsy is feasible, safe, and accurate. This represents the first clinical trial of robotic assistance for MRI-guided transperineal prostate biopsy. The device consists of a robotic needle-guide instrument developed in the investigators Urology Robotics Laboratory. The robot orients a needle-guide on target based on MRI. The physician verifies the alignment and manually takes the biopsy, as usual. Pre-clinical tests showed that the robot operates precisely and safely in the MRI scanner and does not deteriorate imaging quality.

ELIGIBILITY:
Inclusion Criteria:

* men between the ages of 35 and 75,
* have a negative 12 core prostate biopsy, and
* must have one of the following "high risk" features:

  * PSA >= 5.0 ng/ml and Prostate Volume <= 50cc,
  * PSA density >= 0.2ng/ml/cc,
  * Percent Free PSA <=10%,
  * PSA velocity > 0.5 ng/ml/year,
  * High Grade Prostate Intraepithelial Neoplasia on previous biopsy, or Atypia on previous biopsy.

Exclusion Criteria:

* bleeding problems,
* metal implants precluding MRI scanning,
* previous rectal surgery, anal stenosis that precludes endorectal coil insertion,
* patients who cannot tolerate anesthesia or in whom anesthesia is considered high-risk, and
* patients who are unwilling or unable to sign informed consent.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07-25 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Three months
Logged unsuccessful attempts to target prostate | 1 year
Time for device setup, image registration, MRI time, biopsy sampling | 1 year
Score for operation of the device | 1 year
  Score assigned by the engineers on a 1 to 5 scale
Score for image deterioration | 1 year
  Score assigned by radiologist on image quality on a 1 to 5 scale
Quality of the obtained biopsy specimen | 1 year
  Score assigned by the pathologist on a 1-5 scale.
Overall grade of the device and procedure | 1 year
  Grade give by urologist, radiologist and anesthesiologist on a 1-5 scale.

SECONDARY OUTCOMES:
Distance from the collected to planned biopsy core center measured on DICOM | One year
Number of needle trajectory corrections needed for alignment of each biopsy core | 1 year
Number of diagnosed prostate cancers | 1 year
Number of positive/total cores for each patient | 1 year
Correlation of pathology findings with cancer specific region (CSR)s on MRI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Allaf, MD, Principal Investigator — Johns Hopkins University; Mark W Ball, MD, Study Director — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Srimathveeravalli G, Kim C, Petrisor D, Ezell P, Coleman J, Hricak H, Solomon SB, Stoianovici D. MRI-safe robot for targeted transrectal prostate biopsy: animal experiments. BJU Int. 2014 Jun;113(6):977-85. doi: 10.1111/bju.12335. Epub 2013 Dec 2. PMID 24118992
- [Background] Kim C, Chang D, Petrisor D, Chirikjian G, Han M, Stoianovici D. Ultrasound probe and needle-guide calibration for robotic ultrasound scanning and needle targeting. IEEE Trans Biomed Eng. 2013 Jun;60(6):1728-34. doi: 10.1109/TBME.2013.2241430. Epub 2013 Jan 21. PMID 23358940
- [Background] Stoianovici D. Technology advances for prostate biopsy and needle therapies. J Urol. 2012 Oct;188(4):1074-5. doi: 10.1016/j.juro.2012.06.127. Epub 2012 Aug 15. No abstract available. PMID 22901579
- [Background] Bonekamp D, Jacobs MA, El-Khouli R, Stoianovici D, Macura KJ. Advancements in MR imaging of the prostate: from diagnosis to interventions. Radiographics. 2011 May-Jun;31(3):677-703. doi: 10.1148/rg.313105139. PMID 21571651
- [Background] Badaan S, Petrisor D, Kim C, Mozer P, Mazilu D, Gruionu L, Patriciu A, Cleary K, Stoianovici D. Does needle rotation improve lesion targeting? Int J Med Robot. 2011 Jun;7(2):138-47. doi: 10.1002/rcs.381. Epub 2011 Mar 1. PMID 21360796
- [Background] Cunha JA, Hsu IC, Pouliot J, Roach Iii M, Shinohara K, Kurhanewicz J, Reed G, Stoianovici D. Toward adaptive stereotactic robotic brachytherapy for prostate cancer: demonstration of an adaptive workflow incorporating inverse planning and an MR stealth robot. Minim Invasive Ther Allied Technol. 2010 Aug;19(4):189-202. doi: 10.3109/13645706.2010.497000. PMID 20642386
- [Background] Stoianovici D, Song D, Petrisor D, Ursu D, Mazilu D, Muntener M, Schar M, Patriciu A. "MRI Stealth" robot for prostate interventions. Minim Invasive Ther Allied Technol. 2007;16(4):241-8. doi: 10.1080/13645700701520735. PMID 17763098
- [Background] Stoianovici D, Patriciu A, Petrisor D, Mazilu D, Kavoussi L. A New Type of Motor: Pneumatic Step Motor. IEEE ASME Trans Mechatron. 2007 Feb 1;12(1):98-106. doi: 10.1109/TMECH.2006.886258. PMID 21528106
- [Background] Muntener M, Patriciu A, Petrisor D, Mazilu D, Bagga H, Kavoussi L, Cleary K, Stoianovici D. Magnetic resonance imaging compatible robotic system for fully automated brachytherapy seed placement. Urology. 2006 Dec;68(6):1313-7. doi: 10.1016/j.urology.2006.08.1089. PMID 17169653
- [Result] Ball MW, Ross AE, Ghabili K, Kim C, Jun C, Petrisor D, Pan L, Epstein JI, Macura KJ, Stoianovici DS, Allaf ME. Safety and Feasibility of Direct Magnetic Resonance Imaging-guided Transperineal Prostate Biopsy Using a Novel Magnetic Resonance Imaging-safe Robotic Device. Urology. 2017 Nov;109:216-221. doi: 10.1016/j.urology.2017.07.010. Epub 2017 Jul 19. PMID 28735018